CLINICAL TRIAL: NCT05168969
Title: Hyperekplexia in Patients With Loss-of-function CTNNB1 Mutation
Brief Title: Hyperekplexia in Patients With CTNNB1 Mutation
Acronym: CTNNB1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 21CH164; ANSM (Other: 2021-A02047-34)
Record Dates: First submitted 2021-12-10; First posted 2021-12-23 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Hyperekplexia; CTNNB1 Gene Mutation
Keywords: Hyperekplexia; CTNNB1; genetic disorder; psychomotor development; intellectual disability; neurological phenomenon; various visual defects; progressive spastic diplegia
MeSH Terms: conditions — Hyperekplexia; Genetic Diseases, Inborn; Intellectual Disability | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient carrying a CTNNB1 syndrome: Recruitment of subjects with CTNNB1 syndrome will be done through health care providers, but also by contacting families through social media and specialized databases.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The families and health care providers will be invited to fill in a questionnaire related to hyperekplexia (clinical, pharmacological, and genetic data).

SUMMARY:
A few years ago, a new genetic disorder (OMIM # 615075) has been associated with loss-of-function variations in the CTNNB1 gene. The clinical features include a delayed psychomotor development usually leading to severe intellectual disability with or without autistic spectrum disorders, progressive spastic diplegia, and various visual defects. Among over 30 cases described worldwide, 2 were reported with an exaggerated startle response to sudden stimulus corresponding to a very rare neurological phenomenon called hyperekplexia. The investigators also have a 3rd patient carrying a CTNNB1 syndrome associated with hyperekplexia.

DETAILED DESCRIPTION:
Hyperekplexia can impair daily life because the affected person will fall unexpectedly and stiffly, causing repeated head- or body- wounds. It may be treated empirically by various drugs. Hyperekplexia has so far not been associated with CTNNB1 variations.

In this study, we aim to describe the prevalence and clinical characteristics of hyperekplexia in CTNNB1 syndrome carriers, in order to improve diagnosis and thus treatment.

The investigators will recruit CTNNB1 subjects through health care providers and also by contacting the families through dedicated social media and databases. The families and health care providers will be invited to fill in a questionnaire related to hyperekplexia (clinical, pharmacological, and genetic data).

ELIGIBILITY:
Inclusion Criteria:

* Patient carrying a CTNNB1 syndrome showing an exaggerated startle response
* child whose parents have signed a consent form to participate in the study

Exclusion Criteria:

* Absence of molecular diagnosis
* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CTNNB1 subjects
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of hyperekplexia in CTNNB1 subjects | on the day of filling in the questionnaire
  Number of children with hyperekplexia and CTNNB1 syndrome

SECONDARY OUTCOMES:
Clinical features of hyperekplexia | on the day of filling in the questionnaire
  Clinical features (developmental, neurological, and visual disorders) of hyperekplexia in CTNNB1 syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Laure MAZZOLA, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No